CLINICAL TRIAL: NCT01517685
Title: Hallelujah Acres Omega 3 Fat Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallelujah Acres (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 20111700
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Omega 3 Fat Status
Keywords: Eicosapentaenoic acid; EPA; Docosahexaenoic acid; DHA; Omega 3 fat; alpha-linoleic acid; ALA; fish oil; flax seed oil
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flax Oil and then Fish Oil (Experimental): All people in the study will use the flax seed oil and then the fish oil.
  Interventions: Dietary Supplement: Organic flax seed oil; Dietary Supplement: fish oil

INTERVENTIONS:
Dietary Supplement: Organic flax seed oil — 2 tablespoons of organic flax seed oil are eaten daily for 8 weeks.
  Other Names: Flora Flax Oil, organic.
Dietary Supplement: fish oil — 5 grams (1 tsp.) of fish oil is eaten per day for 8 weeks.
  Other Names: Pharmax LLC Finest Pure Fish Oil

SUMMARY:
This research is being done to study the effect of taking flax seed oil and fish oil on blood lipids in vegetarians following the Hallelujah Diet. Omega 3 fats are important to our health and we want to see how effective both flax seed oil and fish oil are in raising your Omega 3 Score (higher is better). The Omega 3 Score is one of many indicators that may show your personal risk of dying suddenly from a heart attack.

DETAILED DESCRIPTION:
This study is being conducted to compare the response of individuals to flax seed oil or fish oil, measured by blood lipids. Especially the amount of the long chain omega 3 polyunsaturated fats EPA and DHA will be tested. An omega 3 score for whole blood will be measured. The omega 3 score is the percent sum of omega 3 fats in the blood.

The hypothesis is that 5 grams of fish oil will increase the amount of EPA and DHA in a person's blood to a protective level, and that 30 grams (2 tablespoons) of flax oil will not change the blood levels of EPA significantly and not change the blood concentrations of DHA at all, even for a person consuming a low omega 6 oil diet and following a vegan diet high in fruits and vegetables.

Most of the testing of flax and fish oil has not been done in vegans. This trial will extend this testing to this subpopulation.

ELIGIBILITY:
Inclusion Criteria:

* Must have followed the Hallelujah Diet (or very similar diet) for at least the last two years,
* Must have stable body weight (not gained or lost more than 5 pounds of weight over the last three months)

Exclusion Criteria:

* Pregnancy (all pregnant women should take fish oil, not flax seed oil)
* Currently using fish oil, or flax seed oil,EPA, DHA, or flax seed oil with added DHA
* Eating more than 2 teaspoons of flax seed per day
* Diabetes (fish oil may affect blood sugar levels)
* Generally poor health

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Omega 3 Score | 8 weeks of supplementation before testing
  A finger prick blood sample is analyzed for fatty acids, including the amount of omega 3 fats in the blood. The Omega 3 Score is the amount of EPA and DHA in whole blood as a percent of fat.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donaldson, PhD, Principal Investigator — Hallelujah Acres
Locations (1):
- Hallelujah Acres Research Office / Laboratory, Zillah, Washington, United States